CLINICAL TRIAL: NCT01615848
Title: Comparison Between Mediterranean Diet and High Protein Diet in Women With Pcos: Randomized Controlled Trial
Brief Title: Comparison Between Mediterranean Diet and High Protein Diet in Women With Polycystic Ovary Syndrome (PCOS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMC12043-20kCTIL
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic Ovary syndrome (PCOS); diet; mediterranean diet; high protein diet
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Diet, High-Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mediterranean diet restricted calorie (Experimental): 1500 k/calories 47-51% carbohydrate 14-17% protein 33-36% fat: 7-7.6% saturated fat 22-30% monounsaturated & polyunsaturated fat
  Interventions: Other: mediterranean diet restricted calorie
- high protein diet, restricted calorie (Experimental): 1500 k/calories 40 % carbohydrate 30% protein 30% fat
  Interventions: Other: high protein diet

INTERVENTIONS:
Other: mediterranean diet restricted calorie — 1500 k/cal 30% fat
  Arms: mediterranean diet restricted calorie
Other: high protein diet — 50 pcos diagnosed women will be assigned to high protein diet for 18 month
  Arms: high protein diet, restricted calorie
Other: mediterranean diet restricted calorie — 50 pcos women will be assigned to 1500 k/cal diet for 18 month
  Arms: mediterranean diet restricted calorie

SUMMARY:
Polycystic ovary syndrome (PCOS) affects 5-10% of women and is the most common endocrine syndrome.PCOS is associated with infertility, risk for obesity and type 2 diabetes. The elevated insulin characteristic of PCOS is likely to play a major role in its symptoms. restricted calorie High protein diet and mediterranean diet may improve insulin sensitivity and therefore lower androgen production in women with pcos women.the purpose of this study is to determine which diet is more effective in improving metabolic and reproductive outcomes.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a heterogeneous syndrome affecting 5-10% of women of reproductive age. It is characterized by elevated circulating insulin, reduced insulin sensitivity, infertility, hyperandrogenism, and a multitude of symptoms that result in a decreased quality of life. The elevated insulin characteristic of PCOS is likely to play a major role in its pathogenesis by reducing insulin sensitivity and stimulating excess androgen production hence causing an hormonal imbalance.

Low calories diets have shown to improve pcos symptoms but the optimal diet for all pcos women is still unknown.

In this study, our purpose is to compare two lowering insulin restricted calories diets in order to find the optimal diet for improving metabolic and endocrin outcomes in pcos women we will also investigate which diet has the best long lasting compliance.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome

Exclusion Criteria:

* Pregnancy
* Lactation 6 month prior to study
* Known hyperandrogenism
* More then 5 kg weight loss 6 month prior to study
* Imbalance pituitary hormones
* Alcohol or drug abuse
* Chronic disease - kidney/heart/diabetes/lung
* Psychiatric disease
* Drug use accept contraceptive pills

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
improvement in metabolic outcomes of women with pcos | 18 months

SECONDARY OUTCOMES:
improvement in clinical symptoms: acne, hirsutism and menstrual regularity | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam Geva, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Clalit Health Services, Haifa, Israel, Israel